CLINICAL TRIAL: NCT02539485
Title: Heating Precondition of Streamlined Liner of the Pharynx Airway Decrease the Incidence of Sore Throat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Geng guiqi, PhD, Fudan University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 15381538
Record Dates: First submitted 2015-08-28; First posted 2015-09-03 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-08

CONDITIONS: Complication of Artificial Airway

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- heating precondition (Other): The mean maximum sealing pressure, gas leakage, gastric distension, postoperative sore throat and other complication were compared between heating precondition group and control group.
  Interventions: Other: heating precondition

INTERVENTIONS:
Other: heating precondition — The streamlined liner of the pharynx airway (SLIPA) was heated 2 hours before use.

SUMMARY:
The effect of heating precondition of streamlined liner of the pharynx airway (SLIPA) on respiratory mechanics and sore throat was investigated.

ELIGIBILITY:
Inclusion Criteria:

* Hysteroscopic surgery
* General anesthesia

Exclusion Criteria:

* Upper respiratory disease
* Communication disfunction

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | 5 minutes
postoperative sore throat | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Guiqi Geng, PhD, Principal Investigator — obstetric & gynecology hospital
Locations (1):
- Obstetric & Gynecology Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Geng G, Chen Y, Liu H. Preheating of streamlined liner of pharyngeal airway (SLIPA) reduced the related complications: a randomized control study. J Clin Monit Comput. 2017 Jun;31(3):547-550. doi: 10.1007/s10877-016-9875-z. Epub 2016 Apr 8. PMID 27059218